CLINICAL TRIAL: NCT03453268
Title: Impact of Reducing Antihypertensive Treatment on Mortality in Frail Subjects With Low Systolic Blood Pressure (SBP). Multicenter, Randomized Controlled Study of Subjects Aged 80 and Over, Living in Nursing Homes and Other IMS.
Brief Title: Impact of Reducing Antihypertensive Treatment on Mortality in Frail Subjects With Low Systolic Blood Pressure (SBP).
Acronym: RETREAT-FRAIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P160602J; 2017-A01646-47 (Other: IDRCB)
Record Dates: First submitted 2018-01-31; First posted 2018-03-05 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Hypertension
Keywords: Blood pressure; Aged; Frailty; Polypharmacy
MeSH Terms: conditions — Hypertension; Frailty

STUDY DESIGN:
Intervention Model Description: Therapeutic strategies: reduction of the antihypertensive treatment (intervention arm) vs. usual treatment (control arm)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1: Interventional (drug reduction) (Other): STEP DOWN strategy.
  Proposition of reduction of the number of antihypertensive medication according to:
  * the systolic blood pressure levels,
  * co-morbidities
  Interventions: Other: STEP DOWN strategy
- 2: Control (Other): Usual treatment
  Interventions: Other: Control

INTERVENTIONS:
Other: STEP DOWN strategy — reduction of the number of antihypertensive medication according to:
  * the systolic blood pressure levels,
  * co-morbidities
  Arms: 1: Interventional (drug reduction)
Other: Control — usual treatment
  Arms: 2: Control

SUMMARY:
The investigators hypothesize that a gradual reduction in antihypertensive treatment in medical-social institutions patients with low systolic blood pressure (SBP) can improve survival through a controlled increase in SBP and a decrease in secondary morbidity due to 'overmedication'.

Accordingly, the investigators propose a randomized, case/control trial in NH patients ≥ 80 years with a SBP<130 mmHg with >1 anti-Htn drugs. This trial will consist of two parallel arms: the intervention arm will entail antihypertensive drug step-down, while the control arm will comprise the standard anti-hypertensive treatment.

DETAILED DESCRIPTION:
High blood pressure (BP), principally systolic hypertension, is a common condition in older people and is considered a major determinant not only of cardiovascular morbidity and mortality, but also of several other age-related diseases, including frailty, cognitive decline and loss of autonomy. The Hypertension in the Very Elderly Treatment (HYVET) study showed the beneficial effect of antihypertensive treatment in patients ≥ 80 years. More recently, the Systolic Blood Pressure Intervention Trial (SPRINT) study showed that even in subjects 75 years and older, CVD outcomes and total mortality were reduced with intensive treatment as compared to the standard therapeutic strategies. However, both HYVET and SPRINT were conducted in selected populations since they excluded the most frail subjects, those with clinically significant cognitive decline and dementia, those with several cardiovascular and other co-morbidities, as well as patients living in medical-social institutions.

* Interestingly, observational studies in these frail people, have shown no or even an inverse relationship between BP and morbidity and mortality. The PARTAGE longitudinal study was performed in 1130 subjects ≥ 80 years living in medical-social institutions. These subjects were receiving at mean 7.1 drugs/day; 2/3 of them were under antihypertensive drugs (mean 2.2 drugs/day). The PARTAGE study showed an over-mortality in hypertensive subjects with low SBP (<130 mmHg) treated with 2 or more antihypertensive drugs. These individuals, who represented 20% of the total studied population, exhibited 80% increase in mortality compared to all other groups, even after adjustment for several comorbidities.
* The recent European guidelines for hypertension indicate that in people ≥ 80 years with SBP≥160 mmHg there is evidence to recommend reducing SBP to between 150 and 140 mmHg. However, no recommendation exists on which strategy to follow if treatment decreases SBP to lower levels (ex: 120 mmHg) especially on the more frail and polymedicated patients of that age. Thus, in this case, physicians can either continue the same treatment of reduce the number of drugs.
* These contrasting results in old hypertensives reflects the enormous functional heterogeneity among individual of this age-group and clearly show that functional status rather than chronological age should guide therapeutic strategies. Thus, the guidelines for robust older individuals cannot be extrapolated to very old, frail individuals, who have been completely excluded from the above-mentioned clinical trials.

The only way is to conduct a controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 80 and over
* Patients living in nursing homes
* Patients with a SBP < 130 mmHg measured in Medical-Social Institutions using the connected blood pressure monitor supplied for the study (average of the last 2 out of 3 measurements after 10 min rest)
* Hypertensive patients whose treatment contains at least 2 antihypertensive molecules and whose treatment has been stabilised for at least :

  * 3 weeks in the case of the introduction or discontinuation of an anti-HBP drug
  * 2 weeks in the case of a change in the dosage of one of the anti-HBP drugs.
* Patients affiliated to a social security scheme
* Patients who have signed the informed consent form (failing which, the legal representative)
* Patients with dementia or with a severe reduction in physical function (impaired vision, asthenia, advanced osteoarthritis, severe tremors, etc.) and/or cognitive function may be included in this study with the agreement of their carers or family/relatives.

Exclusion Criteria:

* Patients in whom no antihypertensive molecule can be reduced for specific reasons (heart failure with ejection fraction <40%, fluid retention due to heart failure, coronary artery disease and diabetic nephropathy).
* Patients with an estimated life expectancy of <3 months
* Patients who have already been included in this study or in another study at the same time

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1048 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | up to 48 months
  All-cause mortality in each of the two groups during follow-up (maximum 48 months depending on when the patient was included).

SECONDARY OUTCOMES:
Cause of death | up to 48 months
  Occurrence of major CV events (myocardial infarction, hospitalisation for heart failure, stroke, other serious CV complication requiring specific management or hospitalisation)
Blood pressure analysis | up to 48 months
  SBP, diastolic blood pressure (DBP), pulse pressure (PP) and heart rate (HR) in the sitting position (or supine if sitting is not possible) and standing position (if possible), during the 24 to 48 month follow-up period.s
Evaluation of frailty | up to 48 months
  Frailty tests: weight, muscle strength (handgrip), Short Physical Performance Battery (SPPB) and assessment of independence using the ADL (Activities of Daily Living) scale every 6 months during the follow-up period at medical visits.
Evaluation of cognitive function | up to 48 months
  Assessment of cognitive functions by MMSE (Mini Mental State Evaluation) every six months during the follow-up period at medical visits.
Assesment of fall and fractures | up to 48 months
  Number of falls and fractures
Medication assessment | up to 48 months
  Total number of medications: number of antihypertensive medications during the 24 to 48 month follow-up period.
Evaluation of Quality of life | up to 48 months
  Quality of life scales (EQ 5D) once a year during the follow-up period at medical visits.
Onset of cardiac decompensation | up to 48 months
  Occurrence of cardiac decompensation, whether fatal or not, and monitoring of changes in blood pressure.
Patient at high risk of decompensation | up to 48 months
  Number of patients at high risk of cardiac decompensation.

CONTACTS AND LOCATIONS:
Overall Officials: Athanase BENETOS, MD, PhD, Principal Investigator — CHRU NANCY - Pôle Gérontologie
Locations (124):
- France (124):
  - CHU Angoulême (Expert center), Angoulême
  - Font Douce (Nursing Home), Angoulême
  - Keriolet (Nursing Home), Auray
  - Kerleano (Nursing Home), Auray
  - Le Parc de la Plesse (Nursing Home), Avrillé
  - Sentiers d'Automne (Nursing Home), Bains-les-Bains
  - Parisot (Nursing Home), Bainville-sur-Madon
  - EHPAD du CH (Nursing Home), Bar-sur-Seine
  - EHPAD Fontarce (Nursing Home), Bar-sur-Seine
  - USLD du CH (Nursing Home), Bar-sur-Seine
  - Saint Charles (Nursing Home), Bayon
  - Argia (Nursing Home), Bayonne
  - EHPAD du Prisse (Nursing home), Bayonne
  - Goxoki (Nursing Home), Bayonne
  - EHPAD CH de Valence (Nursing home), Beauvallon
  - EHPAD Simone de Beauvoir (Nursing Home), Béziers
  - Espace Perréal (Nursing Home), Béziers
  - USLD Espace Perréal (Nursing Home), Béziers
  - CHU Bordeaux (Expert center), Bordeaux
  - La Croix Du Gue (Nursing Home), Bouguenais
  - Poincaré (Nursing Home), Bouxières-aux-Dames
  - Les Rives d'Ode (Nursing Home), Carcassonne
  - Les jardin de Sophia (Nursing Home), Castelnau-le-Lez
  - EHPAD de Monges (Nursing Home), Castres
  - La Villégiale Saint Jacques (Nursing Home), Castres
  - Saint Martin (Nursing Home), Charmes
  - Saint Jean (Nursing Home), Charmois-l'Orgueilleux
  - EHPAD CH Cotentin Pasteur (Nursing Home), Cherbourg
  - Centre pour Personnes Agées (Nursing Home), Colmar
  - Diaconnat (Nursing home), Colmar
  - Chantereine-Orpea (Nursing Home), Coubron
  - Le Hameau de Saubagnacq (Nursing Home), Dax
  - CHU Dijon (Expert center), Dijon
  - EHPAD CHU Dijon Bourgogne (Nursing Home), Dijon
  - Les Bégonias (Nursing Home), Dijon
  - Les marguerites (Nursing Home), Dijon
  - Port du Canal (Nursing Home), Dijon
  - EHPAD Simone Veil (Nursing Home), Eaubonne
  - Bas-Château (Nursing Home), Essey-lès-Nancy
  - Belfontaine (Nursing Home), Fontaine-lès-Dijon
  - Accueil Vologne (Nursing Home), Granges-sur-Vologne
  - Vallée Don (Nursing Home), Guémené-Penfao
  - EHPAD Orpéa (Nursing home), La Talaudière
  - Baudinet De Courcelles (Nursing home), Lay-Saint-Christophe
  - CHU Lille (Expert center), Lille
  - Les Bateliers (Nursing Home), Lille
  - Saint Antoine de Padoue (Nursing Home), Lille
  - EHPAD de Lormont (Nursing Home), Lormont
  - Sainte Thérèse (Nursing Home), Ludres
  - Saint Charles (Nursing Home), Lunéville
  - CHU Lyon (Expert center), Lyon
  - EHPAD Constant (Nursing Home), Lyon
  - La Renaissance-Orpea (Nursing Home), Marseille
  - Bon repos (Nursing Home), Maxéville
  - Saint Sauveur (Nursing Home), Maxéville
  - Félix Marechal (Nursing Home), Metz
  - USLD Nouvielle (Nursing Home), Mont-de-Marsan
  - Coteaux de Montmorency (Nursing Home), Montmorency
  - Jeanne Callarec (Nursing Home), Montmorency
  - Antonin Balmès (Nursing Home), Montpellier
  - CHU Montpellier (Expert center), Montpellier
  - CSPA Bellevue (Nursing Home), Montpellier
  - EHPAD du CH (Nursing Home), Muret
  - Les Cygnes (Nursing Home), Nancy
  - Notre Maison (Nursing home), Nancy
  - Saint Charles EHPAD (Nursing Home), Nancy
  - Saint Charles USLD (Nursing Home), Nancy
  - Saint Joseph (Nursing Home), Nancy
  - Saint Stanislas (Nursing Home), Nancy
  - Gériatrie - CHRU de Nancy (Expert center), Nancy
  - Beauséjour (Nursing Home), Nantes
  - CHU Nantes (Expert center), Nantes
  - La Chézalière LNA Santé (Nursing Home), Nantes
  - CHU Nice (Expert center), Nice
  - EHPAD Cimiez du CHU (Nursing Home), Nice
  - EHPAD GHAM (Nursing Home), Nogent-sur-Seine
  - Bethel (Nursing Home), Oberhausbergen
  - Les Jardins d'Olonne (Nursing Home), Olonne-sur-Mer
  - Résidence Mer et Estuaire (Nursing Home), Paimboeuf
  - APHP (Expert center), Paris
  - EHPAD Broca (Nursing Home), Paris
  - La Collégiale (Nursing Home), Paris
  - Saint Jacques Orpea (Nursing Home), Paris
  - Trocadéro-Orpéa (Nursing Home), Paris
  - USLD Pessac (Nursing Home), Pessac
  - CHU Périgueux (Expert center), Périgueux
  - EHPAD Parrot (Nursing Home), Périgueux
  - Avant-Garde (Nursing Home), Pompey
  - La Salle (Nursing Home), Pompey
  - Nazareth (Nursing Home), Pont-Sainte-Marie
  - Saint Jean (Nursing Home), Portieux
  - Jacques Mellez (Nursing Home), Raon-l'Étape
  - CHU Reims (Expert center), Reims
  - AHPAD AB2 Wilson (Nursing Home), Reims
  - Résidence Roux CHU Reims (Nursing Home), Reims
  - Julien Monnard (Nursing Home), Romilly-sur-Seine
  - Le Clos des platanes (Nursing Home), Romilly-sur-Seine
  - EHPAD Mer Et Pins (Nursing Home), Saint-Brevin-les-Pins
  - Mer et Pins Fleur d'Ajonc (Nursing Home), Saint-Brevin-les-Pins
  - Mer et Pins les Sylphes (Nursing Home), Saint-Brevin-les-Pins
  - Saint Deodat (Nursing Home), Saint-Dié
  - Fauriel (Nursing Home), Saint-Etienne
  - EHPAD de Saint Genest (Nursing Home), Saint-Genest
  - Udazkena (Nursing Home), Saint-Jean-de-Luz
  - Hotel Club (Nursing Home), Saint-Max
  - EHPAD De Senones (Nursing Home), Senones
  - EHPAD Sézanne (Nursing Home), Sézanne
  - CHU Strasbourg (Expert center), Strasbourg
  - EHPAD Bois Fleuri (Nursing Home), Strasbourg
  - EHPAD CHRU Robertsau (Nursing Home), Strasbourg
  - La Christinière ACPPA (Nursing Home), Taluyers
  - Sainte Sophie (Nursing Home), Thiaucourt-Regniéville
  - CHU Toulouse (Expert center), Toulouse
  - Jolimont Marengo Orpea (Nursing Home), Toulouse
  - Clinique les Minimes (Nursing Home), Toulouse
  - Klarene-Orpea (Nursing Home), Tournan-en-Brie
  - CHP Cotentin Simone Veil (Nursing Home), Valognes
  - EHPAD Maison du Lac (Nursing Home), Vannes
  - USLD Maison du Lac (Nursing Home), Vannes
  - Sainte Catherine (Nursing Home), Verdun
  - Saint Joseph (Nursing Home), Ville-sur-Illon
  - Montagne de Reims (Nursing home), Villers-Allerand
  - Villa Saint-Pierre (Nursing Home), Villers-lès-Nancy
  - Les Buissons (Nursing Home), Xertigny

REFERENCES:
- [Derived] Benetos A, Gautier S, Freminet A, Metz A, Labat C, Georgiopoulos I, Bertin-Hugault F, Beuscart JB, Hanon O, Karcher P, Manckoundia P, Novella JL, Diallo A, Vicaut E, Rossignol P; RETREAT-FRAIL Study Group. Reduction of Antihypertensive Treatment in Nursing Home Residents. N Engl J Med. 2025 Nov 20;393(20):1990-2000. doi: 10.1056/NEJMoa2508157. Epub 2025 Aug 29. PMID 40879421